CLINICAL TRIAL: NCT02065375
Title: A Multicenter, Randomized, Dose-Ranging, Double-Masked, Placebo-Controlled Phase 2 Study Evaluating the Safety and Efficacy of RTA 408 Ophthalmic Suspension for the Treatment of Ocular Inflammation and Pain Following Ocular Surgery
Brief Title: RTA 408 Ophthalmic Suspension for the Treatment of Ocular Inflammation and Pain Following Ocular Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RTA 408-C-1307
Record Dates: First submitted 2014-02-13; First posted 2014-02-19 (Estimated); Results first posted 2023-04-19 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Inflammation and Pain Following Ocular Surgery
Keywords: RTA 408; Ocular surgery; Cataract surgery; Ocular inflammation; Ocular pain; Eye inflammation; omaveloxolone
MeSH Terms: conditions — Inflammation; Eye Pain; Endophthalmitis | interventions — omaveloxolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Omaveloxolone Ophthalmic Suspension 1.0% (Experimental): Patients will receive a single drop of Omaveloxolone Ophthalmic suspension 1.0% instilled into the study eye twice daily (approximately 12 hours apart) for 14 days, beginning 24 ± 6 hours after surgery
  Interventions: Drug: Omaveloxolone Ophthalmic Suspension 1.0%
- Omaveloxolone Ophthalmic Suspension 0.5% (Experimental): Patients will receive a single drop of Omaveloxolone Ophthalmic suspension 0.5% instilled into the study eye twice daily (approximately 12 hours apart) for 14 days, beginning 24 ± 6 hours after surgery
  Interventions: Drug: Omaveloxolone Opthalmic Suspension 0.5%
- Placebo (Placebo Comparator): Patients will receive a single drop of vehicle for Omaveloxolone Ophthalmic suspension was instilled into the study eye twice daily (approximately 12 hours apart) for 14 days, beginning 24 ± 6 hours after surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omaveloxolone Ophthalmic Suspension 1.0%
  Other Names: RTA 408
  Arms: Omaveloxolone Ophthalmic Suspension 1.0%
Drug: Omaveloxolone Opthalmic Suspension 0.5%
  Other Names: RTA 408
  Arms: Omaveloxolone Ophthalmic Suspension 0.5%
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study assesses the efficacy and safety of two concentrations of RTA 408 Ophthalmic Suspension in the treatment of patients who have inflammation and pain following ocular surgery.

DETAILED DESCRIPTION:
Following ophthalmic surgery, the current standard of care includes a topical ophthalmic corticosteroid or other anti-inflammatory agent to treat ocular inflammation and improve patient comfort. If left untreated, inflammation of the eye may result in further ocular complications including scarring, vision loss, or blindness. Although the exact dosing regimen is physician-dependent, patients are typically prescribed a topical corticosteroid for a period of 2-4 weeks following surgery, being tapered over the course of delivery as the inflammation subsides. Topical anti-inflammatory agents are usually administered multiple times per day, particularly in the early period following ophthalmic surgery. Continuing efforts in drug development aim to identify alternatives to ophthalmic corticosteroid use, due to their well-known local and systemic negative side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Be greater than or equal to 18 years of age of either sex or any race;
2. Have undergone unilateral cataract extraction via phacoemulsification on the day prior to study enrollment/randomization;
3. Have a grade of ≥2 in anterior chamber cell score on day after surgery (Day 1);
4. Have a potential post-operative pin-hole visual acuity (VA) of greater than 1.0 logarithm of the minimum angle of resolution (logMAR) in the operative eye and fellow eye as measured using an Early Treatment for Diabetic Retinopathy Study (ETDRS) chart;

Exclusion Criteria:

1. Have any intraocular inflammation present in the study eye during the screening slit lamp examination;
2. Have a score greater than "0" on the Ocular Pain Assessment at Screening in the study eye;
3. Have an immunosuppressive disease or an autoimmune disease that in the opinion of the Investigator could affect the quality of the ocular surface;
4. Have active or chronic/recurrent ocular or systemic disease that is uncontrolled and will likely affect wound healing;
5. Have an intraocular pressure (IOP) ≤ 5 mmHg in either eye;
6. Require the use of a contact lens or a collagen shield within 72 hours of investigational drug treatment or during the study period in the study eye; be unwilling to discontinue use of contact lenses during study period in the study eye;
7. Require use of non-diagnostic topical ophthalmic solutions (other than perioperative mydriatics, anesthetics and antiseptics, prophylactic antibiotics, lid scrubs for mild blepharitis, or artificial tears for the management of dry eye) in the study eye for the duration of the study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2014-02-28 (Actual); Primary Completion 2014-09-30 (Actual); Study Completion 2014-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Garden Grove, California
  - Fort Myers, Florida
  - Kansas City, Missouri
  - Elizabeth City, North Carolina
  - Austin, Texas
  - Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Omaveloxolone Ophthalmic Suspension 1.0%: Patients received a single drop of Omaveloxolone Ophthalmic suspension 1.0% instilled into the study eye twice daily (approximately 12 hours apart) for 14 days, beginning 24 ± 6 hours after surgery
  Omaveloxolone Ophthalmic Suspension 1.0%
- Omaveloxolone Ophthalmic Suspension 0.5%: Patients received a single drop of Omaveloxolone Ophthalmic suspension 0.5% instilled into the study eye twice daily (approximately 12 hours apart) for 14 days, beginning 24 ± 6 hours after surgery
  Omaveloxolone Opthalmic Suspension 0.5%
- Placebo: Patients received a single drop of vehicle for Omaveloxolone Ophthalmic suspension instilled into the study eye twice daily (approximately 12 hours apart) for 14 days, beginning 24 ± 6 hours after surgery
  Placebo
Period: Overall Study
Arm/Group | Omaveloxolone Ophthalmic Suspension 1.0% | Omaveloxolone Ophthalmic Suspension 0.5% | Placebo
Started | 37 | 33 | 39
Completed Treatment | 19 | 15 | 25
Completed | 37 | 33 | 39
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population (all randomized patients with available data)
Groups:
- Total: Total of all reporting groups
Arm/Group | Omaveloxolone Ophthalmic Suspension 1.0% | Omaveloxolone Ophthalmic Suspension 0.5% | Placebo | Total
Number analyzed (Participants) | 37 | 33 | 39 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (9.7) | 68.1 (9.31) | 68.9 (9.47) | 68.3 (9.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 18 | 20 | 61
  Male | 14 | 15 | 19 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 2 | 13
  Not Hispanic or Latino | 30 | 28 | 37 | 95
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 3 | 2 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 6 | 3 | 15
  White | 27 | 24 | 34 | 85
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 37 | 33 | 39 | 109

OUTCOME MEASURES:

1. Primary Outcome: Absence of Anterior Chamber Cells at Day 15 (Visit 5)
Description: Count of participants who had absence of anterior chamber cells at Day 15. White blood cells were counted. In a healthy eye, the anterior chamber should not have any blood cells present. "Yes" indicates an absence of anterior chamber cells. Data for visits after a patient was discontinued for lack of efficacy were imputed as failures and missing data were imputed using last observation carried forward.
Time Frame: 15 days after the participant receives the first dose
Population: Intent-to-treat population (all randomized patients with available data). Data for visits after a patient was discontinued for lack of efficacy were imputed as failures and missing data were imputed using last observation carried forward.
Measure: Count of Participants; unit: Participants
Groups:
- Omaveloxolone Ophthalmic Suspension 1.0%: Patients will receive a single drop of Omaveloxolone Ophthalmic suspension 1.0% instilled into the study eye twice daily (approximately 12 hours apart) for 14 days, beginning 24 ± 6 hours after surgery
  Omaveloxolone Ophthalmic Suspension 1.0%
- Omaveloxolone Ophthalmic Suspension 0.5%: Patients will receive a single drop of Omaveloxolone Ophthalmic suspension 0.5% instilled into the study eye twice daily (approximately 12 hours apart) for 14 days, beginning 24 ± 6 hours after surgery
  Omaveloxolone Opthalmic Suspension 0.5%
- Placebo: Patients will receive a single drop of vehicle for Omaveloxolone Ophthalmic suspension was instilled into the study eye twice daily (approximately 12 hours apart) for 14 days, beginning 24 ± 6 hours after surgery
  Placebo
Arm/Group | Omaveloxolone Ophthalmic Suspension 1.0% | Omaveloxolone Ophthalmic Suspension 0.5% | Placebo
Number analyzed (Participants) | 37 | 33 | 39
Participants
  Yes | 10 | 12 | 11
  No | 27 | 21 | 28
Statistical Analysis 1: Comparison: Omaveloxolone Ophthalmic Suspension 1.0% vs Placebo; Test type: Superiority; p = 0.4543, Chi-squared; p values from Pearson chi-squared statistical test between the Omaveloxolone Ophthalmic suspension 1.0% and placebo were one sided; Difference in proportion of patients = -1.2, 95% CI 2-sided [-21.3 to 18.9]
Statistical Analysis 2: Comparison: Omaveloxolone Ophthalmic Suspension 0.5% vs Placebo; Test type: Superiority; p = 0.2297, Chi-squared; p values from Pearson chi-squared statistical test between the Omaveloxolone Ophthalmic suspension 0.5% and placebo were one sided; Difference in proportion of patients = 8.2, 95% CI 2-sided [-13.5 to 29.8]

2. Primary Outcome: Absence of Ocular Pain at Day 4 (Visit 3)
Description: Participants were asked to report their pain on Day 4 using the Numerical Pain Rating Scale (NPRS) for patients receiving active drug compared to patients receiving placebo. The NPRS is an 11-point numeric scale, which ranges from "0" representing "no pain" to "10" representing the "worst pain imaginable". Lower scores indicate less pain. Participants reporting '0' were recorded as "Yes" while patients reporting any other pain score were recorded as "No". Data for visits after a patient was discontinued for lack of efficacy were imputed as failures and missing data were imputed using last observation carried forward.
Time Frame: 4 days after the participant receives the first dose
Population: Intent-to-treat population (all randomized patients with available data).
Measure: Count of Participants; unit: Participants
Arm/Group | Omaveloxolone Ophthalmic Suspension 1.0% | Omaveloxolone Ophthalmic Suspension 0.5% | Placebo
Number analyzed (Participants) | 37 | 33 | 39
Participants
  Yes | 11 | 9 | 20
  No | 26 | 24 | 19
Statistical Analysis 1: Comparison: Omaveloxolone Ophthalmic Suspension 1.0% vs Placebo; Test type: Superiority; p = .0280, Chi-squared; [statistical method as in outcome 1, analysis 1]; Difference in proportion of patients = -21.6, 95% CI 2-sided [-43.1 to 0.00]
Statistical Analysis 2: Comparison: Omaveloxolone Ophthalmic Suspension 0.5% vs Placebo; Test type: Superiority; p = 0.0192, Chi-squared; [statistical method as in outcome 1, analysis 2]; Difference in proportion of patients = -24.0, 95% CI 2-sided [-45.8 to -2.2]

ADVERSE EVENTS:
Time Frame: From Day 1 (24 +/- 6 hours after surgery) to Day 21
Groups:
- Omaveloxolone Ophthalmic Suspension 1.0%: Study Eye: Patients received a single drop of Omaveloxolone Ophthalmic suspension 1.0% instilled into the study eye twice daily (approximately 12 hours apart) for 14 days, beginning 24 ± 6 hours after surgery.
  This arm describes adverse events in the study eye only.
  Omaveloxolone Ophthalmic Suspension 1.0%
- Omaveloxolone Ophthalmic Suspension 1.0%: Non-study Eye: Patients received a single drop of Omaveloxolone Ophthalmic suspension 1.0% instilled into the study eye twice daily (approximately 12 hours apart) for 14 days, beginning 24 ± 6 hours after surgery.
  This arm describes adverse events in the non-study eye only.
  Omaveloxolone Ophthalmic Suspension 1.0%
- Omaveloxolone Ophthalmic Suspension 0.5%: Study Eye: Patients received a single drop of Omaveloxolone Ophthalmic suspension 0.5% instilled into the study eye twice daily (approximately 12 hours apart) for 14 days, beginning 24 ± 6 hours after surgery
  This arm describes adverse events in the study eye only.
  Omaveloxolone Ophthalmic Suspension 0.5%
- Omaveloxolone Ophthalmic Suspension 0.5%: Non-study Eye: Patients received a single drop of Omaveloxolone Ophthalmic suspension 0.5% instilled into the study eye twice daily (approximately 12 hours apart) for 14 days, beginning 24 ± 6 hours after surgery
  This arm describes adverse events in the non-study eye only.
  Omaveloxolone Ophthalmic Suspension 0.5%
- Placebo: Study Eye: Patients received a single drop of vehicle for Omaveloxolone Ophthalmic suspension instilled into the study eye twice daily (approximately 12 hours apart) for 14 days, beginning 24 ± 6 hours after surgery
  This arm describes adverse events in the study eye only.
  Placebo
- Placebo: Non-study Eye: Patients received a single drop of vehicle for Omaveloxolone Ophthalmic suspension instilled into the study eye twice daily (approximately 12 hours apart) for 14 days, beginning 24 ± 6 hours after surgery
  This arm describes adverse events in the non-study eye only.
  Placebo
- Omaveloxolone Ophthalmic Suspension 1.0%: Non-ocular AE: Patients received a single drop of Omaveloxolone Ophthalmic suspension 1.0% instilled into the study eye twice daily (approximately 12 hours apart) for 14 days, beginning 24 ± 6 hours after surgery
  This arm describes non-ocular adverse events only.
  Omaveloxolone Ophthalmic Suspension 1.0%
- Omaveloxolone Ophthalmic Suspension 0.5%: Non-ocular AE: Patients received a single drop of Omaveloxolone Ophthalmic suspension 0.5% instilled into the study eye twice daily (approximately 12 hours apart) for 14 days, beginning 24 ± 6 hours after surgery
  This arm describes non-ocular adverse events only.
  Omaveloxolone Ophthalmic Suspension 0.5%
- Placebo: Non-ocular AE: Patients received a single drop of vehicle for Omaveloxolone Ophthalmic suspension instilled into the study eye twice daily (approximately 12 hours apart) for 14 days, beginning 24 ± 6 hours after surgery
  This arm describes non-ocular adverse events only.
  Placebo
Arm/Group | Omaveloxolone Ophthalmic Suspension 1.0%: Study Eye | Omaveloxolone Ophthalmic Suspension 1.0%: Non-study Eye | Omaveloxolone Ophthalmic Suspension 0.5%: Study Eye | Omaveloxolone Ophthalmic Suspension 0.5%: Non-study Eye | Placebo: Study Eye | Placebo: Non-study Eye | Omaveloxolone Ophthalmic Suspension 1.0%: Non-ocular AE | Omaveloxolone Ophthalmic Suspension 0.5%: Non-ocular AE | Placebo: Non-ocular AE
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/37 | 0/33 | 0/33 | 0/39 | 0/39 | 0/37 | 0/33 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37 | 0/33 | 0/33 | 0/39 | 0/39 | 0/37 | 0/33 | 0/39
Other Adverse Events (participants affected / at risk) | 18/37 | 0/37 | 15/33 | 2/33 | 13/39 | 1/39 | 2/37 | 2/33 | 1/39
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omaveloxolone Ophthalmic Suspension 1.0%: Study Eye (N=37) | Omaveloxolone Ophthalmic Suspension 1.0%: Non-study Eye (N=37) | Omaveloxolone Ophthalmic Suspension 0.5%: Study Eye (N=33) | Omaveloxolone Ophthalmic Suspension 0.5%: Non-study Eye (N=33) | Placebo: Study Eye (N=39) | Placebo: Non-study Eye (N=39) | Omaveloxolone Ophthalmic Suspension 1.0%: Non-ocular AE (N=37) | Omaveloxolone Ophthalmic Suspension 0.5%: Non-ocular AE (N=33) | Placebo: Non-ocular AE (N=39)
Anterior chamber pigmentation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ciliary hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 11 (11) | 0 (0) | 9 (10) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal deposits (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal disorder (Eye disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal oedema (Eye disorders) | 3 (3) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal pigmentation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal striae (Eye disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystoid macular oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foreign body sensation in eyes (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lenticular opacities (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular discomfort (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 2 (2) | 0 (0) | 3 (4) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Instillation site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2014-02-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT02065375/Prot_000.pdf
  • Statistical Analysis Plan (2014-02-13): https://cdn.clinicaltrials.gov/large-docs/75/NCT02065375/SAP_001.pdf